CLINICAL TRIAL: NCT02933411
Title: Genotypic and Phenotypic Analysis of Adolescents With Heavy Menstrual Bleeding and Low Von Willebrand Activity
Brief Title: Low VW Activity in Adolescent HMB
Acronym: Low VWF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Sarah Sartain, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-39295 LOW VWF
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Von Willebrand Factor Deficiency
Keywords: Bleeding Disorders; Heavy Menstrual Bleeding
MeSH Terms: conditions — Von willebrand factor, deficiency; Hemostatic Disorders; Menorrhagia | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be drawn to assess the number of participants enrolled that have heavy menstrual bleeding and low von willebrand activity disease causing sequence variation in the von willebrand factor gene and other genes affecting bleeding, clotting and blood vessel biology.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: Adolescent women with heavy menstrual bleeding and low von willebrand factor activity.
  Interventions: Other: Genetic Analysis; Other: Medical Record Data Abstraction; Other: Pictorial Blood Assessment Chart (PBAC) score; Other: Complete Bleeding Symptom ISTH Bleeding Assessment Tool

INTERVENTIONS:
Other: Genetic Analysis — Blood sample will be drawn to assess the number of participants enrolled that have sequence variation in the von willebrand factor gene and other genes affecting bleeding, clotting and blood vessel biology.
Other: Medical Record Data Abstraction — The subject's response to intranasal or intravenous desmopressin (DDAVP) challenge performed as part of standard of care will be recorded. The desmopressin is a drug that increases the clotting factor in blood to prevent bleeding.
  Medical and family history including and not limited to age, diagnoses, race/ethnicity, lab values, HMB and low VWF activity diagnoses, and treatment history and outcome will also be recorded.
Other: Pictorial Blood Assessment Chart (PBAC) score — PBAC is a pictorial tool to assess menstrual blood loss. Study team will complete the PBAC assessment with each study participant evaluating and measure response to different treatments for menstrual blood loss in the clinic setting between those with VWD versus other bleeding disorders.
  Other Names: PBAC Score
Other: Complete Bleeding Symptom ISTH Bleeding Assessment Tool — Study participants will complete the ISTH BAT assessment. The ISTH BAT is a questionnaire to aid in the standardized evaluation of the presence and severity of bleeding symptoms.
  Other Names: ISTH BAT Assessment

SUMMARY:
This is a research study for patients diagnosed with heavy menstrual bleeding (HMB) and low Von Willebrand Factor (VWF). Menstruation, also known as a period, is the regular discharge of blood and tissues from the uterus. HMB is having a heavier amount of discharge during menstrual period. Low Von Willebrand Factor means that the participant has lower level of a blood protein that is important for clotting of blood and so, the participant is at a higher risk for bleeding.

The purpose of this project is to study the genetic differences of adolescent females with HMB and low VWF activity and compare the genetic differences with their bleeding manifestations, response to medications and outcome.

DETAILED DESCRIPTION:
One hundred and twenty subjects will be enrolled. Adolescent females with heavy menstrual bleeding (HMB) and low Von Willebrand Factor (VWF) will be recruited.

Data collection will occur from participant's medical records in regards to their low VWF activity and HMB medical history.

Participants will be asked to complete symptom questionnaires in regards to their HMB.

A blood sample will be collected to analyze how many participants have the disease causing sequence variation in the VWF gene and other genes affecting bleeding, clotting and blood vessel biology and correlated with their bleeding history.

The blood sample will be deidentified and stored indefinitely for future research.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarchal females less than 21 years of age
* HMB defined as PBAC score greater than 100
* VWF:Activity more than or equal to 30 and less than or equal to 50 IU/dL x 2
* VWF: Activity /VWF:Ag ratio greater than or equal to 0.6
* Normal VW multimers, if performed

Exclusion Criteria:

* Post menarchal females age greater than or equal to 21 years
* VWF: Activity less than 30 or greater than 50 IU/dL consistently, type 2 or type 3 VWD
* Presence of other bleeding disorders (thrombocytopenia, platelet function defect, coagulation factor deficiency, fibrinogen defect or deficiency)

Max Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Females under the age of 21 years old with heavy menstrual bleeding and low von willebrand factor
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of adolescents with Low VWF and HMB with genetic variations in VWF gene and other genes affecting bleeding, clotting and blood vessel biology | 3 years
  The genetic variations of adolescent females with heavy menstrual bleeding and low von Willebrand factor activity in VWF gene and other genes affecting bleeding, clotting and blood vessel biology

SECONDARY OUTCOMES:
Number of adolescents with Low VWF and HMB with genetic variations and bleeding phenotype (including PBAC score and ISTH-BAT score, response to DDAVP challenge, HMB therapy) | 3 years
  The correlation of subjects with and without genetic variations with bleeding phenotype (including PBAC score, ISTH BAT score, response to DDAVP challenge and HMB therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sartain, MD, Principal Investigator — Texas Children's Hospital, an affiliate of Baylor College of Medicine
Locations (12):
- United States (12):
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Michigan State University, East Lansing, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Joseph M Sanzari Children's Hospital, Hackensack, New Jersey
  - Hemophilia Center of Western New York, Buffalo, New York
  - Mary M. Gooley Hemophilia Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center- Children's Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No